CLINICAL TRIAL: NCT00216580
Title: An Open-label Trial of Risperidone Long-acting Injectable in the Treatment of Subjects With Recent Onset Psychosis
Brief Title: A Pilot Study of the Use of Risperidone Long Acting Injectable in the Treatment of Patients With Recent Onset Psychosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR003358; RIS-PSY-301 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Intramuscular injection; Antipsychotic agents; Long-acting risperidone; Schizophreniform disorders; Schizoaffective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Risperidone, long-acting injectable (Experimental)
  Interventions: Drug: Risperidone, long-acting injectable

INTERVENTIONS:
Drug: Risperidone, long-acting injectable

SUMMARY:
The purpose of the study is to assess the effectiveness and safety of long-acting injectable risperidone in the treatment of patients in the early stage of psychosis

DETAILED DESCRIPTION:
Although many schizophrenia patients currently take oral antipsychotic medications, it is estimated that up to 75% of them have difficulty adhering to the daily oral regimen. Long-acting injectable formulations may eliminate the need for daily medication and enhance patient compliance with the treatment regimen. This study is a pilot project to demonstrate that long-acting risperidone can be used safely and effectively in treating patients in the early stage of psychosis. It is an open-label, single-arm study in patients with recent onset of schizophrenia, schizophreniform disorder, or schizoaffective disorder. There are 3 phases: Wash-out Phase of 7 days, during which current psychotropic medications are discontinued; Oral Treatment Phase, beginning 1 week before the first injection and continuing 3 weeks thereafter, during which risperidone tablets are taken; and Long-Acting Injectable Treatment Phase, during which injections are given every 2 weeks for 24 months. Assessments of effectiveness include Positive and Negative Syndrome Scale (PANSS), a scale for the measurement of symptoms of schizophrenia; time from initiation of treatment to relapse; Calgary Depression Scale for Schizophrenia (CDSS), which assesses symptoms of major depressive disorder in patients with schizophrenia; and Clinical Global Impression (CGI) scales. Safety assessments include the incidence of adverse events and Extrapyramidal Symptom Rating Scale (ESRS) scores throughout the study; clinical laboratory tests (hematology and chemistry) and vital signs (pulse, blood pressure, temperature) at stated intervals. Risperidone oral tablets once daily (1 milligram[mg], 2mg, or 3mg [maximum]) from 1 week before first injection through 3 wks after. Risperidone injections (25mg, 37.5mg, or 50mg [max]) every 2 weeks for 24 months. Doses may be increased or decreased at investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria of the Diagnostic and Statistical Manual of Mental Diseases, 4th edition (DSM-IV) for schizophreniform disorder, schizophrenia, or schizoaffective disorder for no longer than 12 months, and with not more than two hospitalizations for psychosis
* patients who have, during their lifetime, been exposed to a maximum of 12 weeks of antipsychotic medication
* patients who will require at least 12 months of treatment

Exclusion Criteria:

* DSM-IV axis I diagnosis other than schizophreniform disorder, schizophrenia, or schizoaffective disorder
* patients requiring treatment with mood stabilizers or antidepressants at study initiation
* alcohol or drug abuse or dependence, according to DSM-IV criteria
* history of drug allergy, drug hypersensitivity (including risperidone), or neuroleptic malignant syndrome, a rare psychotropic-drug reaction, which may be characterized by confusion, reduced consciousness, high fever or pronounced muscle stiffness
* previous treatment with an injectable antipsychotic medication
* pregnant or nursing females, or those lacking adequate contraception

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2004-02; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Syndrome Scale (PANSS) from baseline to end of study

SECONDARY OUTCOMES:
Time from initiation of treatment to relapse; changes in Calgary Depression Scale for Schizophrenia (CDSS), Clinical Global Impression (CGI) scales, Extrapyramidal Symptom Rating Scale (ESRS) at intervals throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.

REFERENCES:
- See also: An open-label trial of risperidone long-acting injectable in the treatment of subjects with recent onset psychosis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=384&filename=CR003358_CSR.pdf